CLINICAL TRIAL: NCT01177774
Title: Predictive Biomarkers of Conversion to Tourette Syndrome in Children With New-Onset Tics
Brief Title: Assessment of Children With Tic Onset in the Past 6 Months
Acronym: NewTics
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kevin J. Black, M.D., Professor, Washington University School of Medicine
Other Study IDs: 09-1700; K24MH087913 (NIH)
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Tourette Syndrome; Tourette's Disorder; Chronic Motor or Vocal Tic Disorder; Transient Tic Disorder; Tic Disorders; Provisional Tic Disorder
Keywords: functional connectivity MRI; brain volumetry; negative reinforcement; OCD; ADHD
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Recent-onset tics that will persist: Children between 5 to 10 years of age with recent-onset tics (first tic occurred within the past 9 months) who, when reassessed at 1 year after the first tic began (i.e. 6-12 months after study enrollment) will turn out to meet criteria for a chronic tic disorder (including Tourette syndrome). Scheduled follow-up visits will include children over age 10 (initially enrolled at age 5-10).
- Recent-onset tics that will remit: Children between 5 to 10 years of age with recent-onset tics (first tic occurred within the past 9 months) who will no longer have tics when reassessed 1 year after the first tic began (6 to 12 months after study enrollment). Scheduled follow-up visits will include children over age 10 (initially enrolled at age 5-10).
- Tic-free control subjects: Children with no current or past tic disorder of similar age, sex and handedness as the children in the recent-onset tics groups.
- Existing TS/CTD: Children with current tics whose first tics were more than 12 months ago (DSM-5 Tourette's Disorder or Persistent [Chronic] Motor or Phonic Tic Disorder), of similar age, sex and handedness as the children in the recent-onset tics groups.

SUMMARY:
The purpose of this research is to study why most children who have tics never develop Tourette syndrome but some do. In other words, we aim to find features that may predict whose tics will go away and whose tics will continue or worsen, in children ages 5 through 10 years whose first tic occurred within the past 9 months.

DETAILED DESCRIPTION:
Up to 30% of all children will have a tic at some point. However, tics that last a whole year (or more) occur in only 3% of the population. Thus tic persistence may be more unusual than tic onset, yet almost no data exist on which people with recent-onset tics go on to be diagnosable with Tourette syndrome or chronic tic disorder, versus those whose tics are only transient.

The overall goal of this research is to identify, prospectively, what imaging, clinical or neuropsychological features of children who just recently started ticcing will go on to develop a chronic tic disorder (including Tourette syndrome). Hypotheses are derived primarily from studies of patients with established tic disorders.

Aim 1. Study pathophysiology of recent-onset tics. Aim 1a. Identify clinical, neuropsychological, and brain imaging features that differentiate children with recent tic onset ("New Tics" group) from tic-free controls. We will test a priori hypotheses including tic suppression, inattentiveness, caudate nucleus volume, tic severity, and premonitory urges (see "Summary of hypotheses" on the 3rd page of Research Strategy). Secondary analyses will apply support vector machine (SVM) learning to a rich set of data to discover novel, multivariate differences in the New Tics group [3,45]. These data will also include tic phenomenology, psychiatric diagnosis, habit learning, motor dexterity, structural MRI, perfusion MRI, and resting state functional connectivity fMRI (rs-fcMRI).

Aim 1b. Compare New Tics subjects to a group of children who are matched for age but have already had tics for ≥1 year ("Existing TS/CTD"). Since both groups have tics, this comparison will highlight abnormalities that cannot be explained by the mere current presence of tics, including markers of chronicity or adaptation.

Aim 2. Prospective study of tic remission. We will re-evaluate New Tics subjects at the 1-year anniversary of tic onset (the accepted duration criterion for diagnosis of TS/CTD). Our pilot data show good variability in the change in tic symptom severity (i.e., change in YGTSS total tic score from baseline to followup: ΔTTS), so ΔTTS will be the primary dependent variable. We focus on outcome as a continuous variable because no reliable estimate exists for how many New Tics subjects will remit versus go on to diagnosis with TS/CTD. Remission rate also depends on definition and on the thoroughness of the follow-up evaluation [4].

Aim 2a. Study the physiology of tic remission by identifying changes in clinical, neuropsychological, and brain imaging variables that correlate with changes in clinical tic severity (ΔTTS). This Aim benefits from prospective observation and within-subject comparisons. The primary analysis will focus on any markers identified in Aim 1. A secondary analysis will apply machine learning methods for a data-driven approach (support vector regression: SVR).

Aim 2b. Identify predictors of improvement or worsening, i.e. clinical, neuropsychological, and brain imaging features at study entry that correlate significantly with ΔTTS. The 2 primary analyses will relate clinical outcome (ΔTTS) to tic suppression ability and caudate volume at study entry. Secondary analyses will examine other predictors using an SVR machine learning approach.

ELIGIBILITY:
** All subjects **

Inclusion Criteria:

* Age 5-10
* Informed consent from a parent and assent from the child.

  * New Tics Group **

Inclusion Criteria:

* tics now, but developed them only in the past 9 months.

Exclusion criteria: secondary tics, another neurological disorder (not counting migraine), structural brain disease, severe systemic illness, nonproficiency in the English language, and psychiatric illness including mental retardation, autism, substance dependence, current substance abuse, primary psychotic illness, bipolar disorder and current major depression. Psychoactive medications are allowed if their dose has not changed in the past month.

** Existing TS/CTD control group **

Inclusion criteria:

* children who meet DSM-5 criteria for Tourette's Disorder or Persistent Tic Disorder at enrollment
* matched to children from the New Tics group on age (within 1 year), sex, handedness, and ADHD status.

Exclusion criteria: same as for the New Tics group.

** Tic-free controls **

Inclusion criteria: tic-free children matched to children from the New Tics group on age (within 1 year), sex, handedness, and ADHD status.

Exclusion criteria: current or past tic disorder in the subject or a first-degree relative, plus the exclusions listed for the New Tics group.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1. A convenience sample of children age 5-10 who have tics now but whose first-ever tic occurred within the past 9 months. Subjects will be a convenience sample from community and clinical sources.
  2. A control group who already meets criteria for a diagnosis of a chronic tic disorder, matched for age, sex, handedness, and ADHD
  3. A control group who has no tics, matched for age, sex, handedness, and ADHD
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2010-08; Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
DSM-5 diagnosis of a chronic tic disorder at 12 months | 1 year after the onset of tics (6-12 months after the first study visit)
  Research diagnosis of a chronic tic disorder at 12 months (cases), versus those whose tics are absent at 12 months (controls), will define two groups who will be compared on their baseline status (almost a year earlier) on a quantitative measure of functional connectivity maturity, pre-tic BOLD signal, caudate nucleus volume, and several clinical and neuropsychological measures.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J. Black, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, Movement Disorder Clinic, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Beginning in June, 2017, all data other than PHI will follow the NIMH RDoC data sharing policy.
Time Frame: Subject-level data: first data upload approximately 25 September 2018, then twice yearly through the end of the grant period.
Access Criteria: open
URL: https://ndar.nih.gov/edit_collection.html?id=2692

REFERENCES:
- See also: Click here for more information about this study: Predictive Biomarkers of Conversion to Tourette Syndrome in Children with New-Onset Tics — http://www.newtics.info
- See also: Click here for more information about this study: Predictive Biomarkers of Conversion to Tourette Syndrome in Children with New-Onset Tics — http://www.newtics.org
- See also: Tourette Syndrome resources — https://sites.wustl.edu/tics/resources/